CLINICAL TRIAL: NCT02852499
Title: SEPAGES : Following of Atmospheric Pollution Exposure During Pregnancy and Effects on Health
Brief Title: Following of Atmospheric Pollution Exposure During Pregnancy and Effects on Health
Acronym: SEPAGES-1337
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 38RC13.579
Record Dates: First submitted 2016-05-26; First posted 2016-08-02 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteer
Keywords: environmental epidemiology; cohort; atmospheric pollutant; chemical pollutant; growth, neuro-development, respiratory health; big data; biological samples (RNA, DNA, urines ...); e-dohad and exposome
MeSH Terms: interventions — DNER protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mothers: Pregnant women.
  Interventions: Other: Urine sampling; Other: Carry a GPS and BET; Other: Carry pollution sensor; Other: Sampling at the maternity; Other: Self-questionnaires
- Fathers: Futur fathers.
  Interventions: Other: Urine sampling; Other: Self-questionnaires
- Children: Children after childbirth.
  Interventions: Other: Sampling in partum period

INTERVENTIONS:
Other: Urine sampling
  Groups: Fathers; Mothers
Other: Carry a GPS and BET
  Groups: Mothers
Other: Carry pollution sensor
  Groups: Mothers
Other: Sampling at the maternity
  Groups: Mothers
Other: Self-questionnaires
  Groups: Fathers; Mothers
Other: Sampling in partum period — Meconium and a strand of hair.
  Groups: Children

SUMMARY:
The SEPAGES couple-child cohort is coordinated by an Inserm (French National Institute of Health and Medical Research) team of environmental epidemiology. SEPAGES cohort is based on the general population and aims to cover several areas of environmental health research, including endocrine disruptors and air pollutants.

The main objectives is to quantify the impact of pollution during pregnancy and the first years of life on three main health outcomes : growth, respiratory health and neuro-development ; and to better understand the biological mechanism (such as genetic analysis to study the role of environmental factors on genes expression as well as the role of genetic factors on health). The objective is to include 500 families.

DETAILED DESCRIPTION:
SEPAGES is a new type of longitudinal couple-child cohort with repeated clinical examinations during pregnancy and childhood, extensive collection of repeated biological samples from both parents and the child, use of new technologies to assess exposure to air pollution (GPS, personal dosimeter etc.) Throughout the study (during pregnancy and the first years of the child's life), clinical examination and many biological tests (urine, blood, hair) are performed. Exposure to different environmental factors are made several times during pregnancy and the first years of the child's life thanks to personal dosimeters, GPS and accelerometers. During labor and childbirth a number of samples are taken (placenta, tissues, blood, urines, hair, meconium and breast milk). Finally, during the study a number of evaluation questionnaires are given to volunteers via a computer platform in order to have a better understanding of the environment in which they are living.

The SEPAGES cohort follows the rule of the biomedical research. Informed consents are signed by both the father and the mother during the inclusion visit which takes place in the hospital. All ethical and data privacy agreements had been obtained : a favorable opinion was issued by the Comité de Protection des Personnes (CPP) on November 13th, 201 and by the CCTIRS (Comité Consultatif sur le Traitement de l'Information en matière de Recherche dans le domaine de la Santé) on January 09th, 2014. The study was authorised by the Agence Nationale de Sécurité du Médicament(ANSM), on Decmber 17th, 2013 and by the Comité Nationale de l'Informatique et des Libertés (CNIL) on June 26th, 2014.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* < 19 gestational weeks
* > 18 years old
* living in the area of Grenoble
* planning to give birth in one of the four maternities located in Grenoble

Exclusion Criteria:

* not speaking French
* no access to the French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women before 19 getsationel week, older than 18 years old Father of the children Children at birth
Sampling Method: Non-Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2014-07; Primary Completion 2018-02 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Clinical exam : biological sampling | Up to one hour
  Sampling of : meconium, strands of hair, mouth cells, nose cells and a skin test in g
Clinical exam : biological sampling | Up to one hour
  Sampling of : urines, blood in mL

CONTACTS AND LOCATIONS:
Overall Officials: iSABELLE Pin, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Hopital Couple Enfant - Grenoble, La Tronche, France

REFERENCES:
- [Background] Barker DJ, Osmond C, Golding J, Kuh D, Wadsworth ME. Growth in utero, blood pressure in childhood and adult life, and mortality from cardiovascular disease. BMJ. 1989 Mar 4;298(6673):564-7. doi: 10.1136/bmj.298.6673.564. PMID 2495113
- [Background] Barker DJ, Winter PD, Osmond C, Margetts B, Simmonds SJ. Weight in infancy and death from ischaemic heart disease. Lancet. 1989 Sep 9;2(8663):577-80. doi: 10.1016/s0140-6736(89)90710-1. PMID 2570282
- [Background] Barker DJ. The developmental origins of adult disease. J Am Coll Nutr. 2004 Dec;23(6 Suppl):588S-595S. doi: 10.1080/07315724.2004.10719428. PMID 15640511
- [Background] Lawlor DA, Ebrahim S, Davey Smith G. Association of birth weight with adult lung function: findings from the British Women's Heart and Health Study and a meta-analysis. Thorax. 2005 Oct;60(10):851-8. doi: 10.1136/thx.2005.042408. Epub 2005 Jul 29. PMID 16055617
- [Background] Rona RJ, Gulliford MC, Chinn S. Effects of prematurity and intrauterine growth on respiratory health and lung function in childhood. BMJ. 1993 Mar 27;306(6881):817-20. doi: 10.1136/bmj.306.6881.817. PMID 8490372
- [Background] Martinez FD, Wright AL, Taussig LM, Holberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med. 1995 Jan 19;332(3):133-8. doi: 10.1056/NEJM199501193320301. PMID 7800004
- [Background] Haland G, Carlsen KC, Sandvik L, Devulapalli CS, Munthe-Kaas MC, Pettersen M, Carlsen KH; ORAACLE. Reduced lung function at birth and the risk of asthma at 10 years of age. N Engl J Med. 2006 Oct 19;355(16):1682-9. doi: 10.1056/NEJMoa052885. PMID 17050892
- [Background] Stern DA, Morgan WJ, Wright AL, Guerra S, Martinez FD. Poor airway function in early infancy and lung function by age 22 years: a non-selective longitudinal cohort study. Lancet. 2007 Sep 1;370(9589):758-64. doi: 10.1016/S0140-6736(07)61379-8. PMID 17765525
- [Background] Jensen TK, Jorgensen N, Punab M, Haugen TB, Suominen J, Zilaitiene B, Horte A, Andersen AG, Carlsen E, Magnus O, Matulevicius V, Nermoen I, Vierula M, Keiding N, Toppari J, Skakkebaek NE. Association of in utero exposure to maternal smoking with reduced semen quality and testis size in adulthood: a cross-sectional study of 1,770 young men from the general population in five European countries. Am J Epidemiol. 2004 Jan 1;159(1):49-58. doi: 10.1093/aje/kwh002. PMID 14693659
- [Background] Moshammer H, Hoek G, Luttmann-Gibson H, Neuberger MA, Antova T, Gehring U, Hruba F, Pattenden S, Rudnai P, Slachtova H, Zlotkowska R, Fletcher T. Parental smoking and lung function in children: an international study. Am J Respir Crit Care Med. 2006 Jun 1;173(11):1255-63. doi: 10.1164/rccm.200510-1552OC. Epub 2006 Feb 16. PMID 16484675
- [Background] McKeever TM, Lewis SA, Smith C, Collins J, Heatlie H, Frischer M, Hubbard R. Early exposure to infections and antibiotics and the incidence of allergic disease: a birth cohort study with the West Midlands General Practice Research Database. J Allergy Clin Immunol. 2002 Jan;109(1):43-50. doi: 10.1067/mai.2002.121016. PMID 11799364
- [Background] Li YF, Langholz B, Salam MT, Gilliland FD. Maternal and grandmaternal smoking patterns are associated with early childhood asthma. Chest. 2005 Apr;127(4):1232-41. doi: 10.1378/chest.127.4.1232. PMID 15821200
- [Background] Shaheen SO, Sterne JA, Montgomery SM, Azima H. Birth weight, body mass index and asthma in young adults. Thorax. 1999 May;54(5):396-402. doi: 10.1136/thx.54.5.396. PMID 10212102
- [Background] Miller RL, Ho SM. Environmental epigenetics and asthma: current concepts and call for studies. Am J Respir Crit Care Med. 2008 Mar 15;177(6):567-73. doi: 10.1164/rccm.200710-1511PP. Epub 2008 Jan 10. PMID 18187692
- [Background] Breton CV, Byun HM, Wenten M, Pan F, Yang A, Gilliland FD. Prenatal tobacco smoke exposure affects global and gene-specific DNA methylation. Am J Respir Crit Care Med. 2009 Sep 1;180(5):462-7. doi: 10.1164/rccm.200901-0135OC. Epub 2009 Jun 4. PMID 19498054
- [Background] Shaheen SO, Adcock IM. The developmental origins of asthma: does epigenetics hold the key? Am J Respir Crit Care Med. 2009 Oct 15;180(8):690-1. doi: 10.1164/rccm.200906-0893ED. No abstract available. PMID 19824169
- [Background] Foley DL, Craig JM, Morley R, Olsson CA, Dwyer T, Smith K, Saffery R. Prospects for epigenetic epidemiology. Am J Epidemiol. 2009 Feb 15;169(4):389-400. doi: 10.1093/aje/kwn380. Epub 2009 Jan 12. PMID 19139055
- [Background] Baccarelli A, Wright RO, Bollati V, Tarantini L, Litonjua AA, Suh HH, Zanobetti A, Sparrow D, Vokonas PS, Schwartz J. Rapid DNA methylation changes after exposure to traffic particles. Am J Respir Crit Care Med. 2009 Apr 1;179(7):572-8. doi: 10.1164/rccm.200807-1097OC. Epub 2009 Jan 8. PMID 19136372
- [Background] Braback L, Forsberg B. Does traffic exhaust contribute to the development of asthma and allergic sensitization in children: findings from recent cohort studies. Environ Health. 2009 Apr 16;8:17. doi: 10.1186/1476-069X-8-17. PMID 19371435
- [Background] Brauer M, Hoek G, Smit HA, de Jongste JC, Gerritsen J, Postma DS, Kerkhof M, Brunekreef B. Air pollution and development of asthma, allergy and infections in a birth cohort. Eur Respir J. 2007 May;29(5):879-88. doi: 10.1183/09031936.00083406. Epub 2007 Jan 24. PMID 17251230
- [Background] Mortimer K, Neugebauer R, Lurmann F, Alcorn S, Balmes J, Tager I. Air pollution and pulmonary function in asthmatic children: effects of prenatal and lifetime exposures. Epidemiology. 2008 Jul;19(4):550-7; discussion 561-2. doi: 10.1097/EDE.0b013e31816a9dcb. PMID 18520616
- [Background] Pinkerton KE, Joad JP. Influence of air pollution on respiratory health during perinatal development. Clin Exp Pharmacol Physiol. 2006 Mar;33(3):269-72. doi: 10.1111/j.1440-1681.2006.04357.x. PMID 16487273
- [Background] Ritz B, Yu F. The effect of ambient carbon monoxide on low birth weight among children born in southern California between 1989 and 1993. Environ Health Perspect. 1999 Jan;107(1):17-25. doi: 10.1289/ehp.9910717. PMID 9872713
- [Background] Slama R, Darrow L, Parker J, Woodruff TJ, Strickland M, Nieuwenhuijsen M, Glinianaia S, Hoggatt KJ, Kannan S, Hurley F, Kalinka J, Sram R, Brauer M, Wilhelm M, Heinrich J, Ritz B. Meeting report: atmospheric pollution and human reproduction. Environ Health Perspect. 2008 Jun;116(6):791-8. doi: 10.1289/ehp.11074. PMID 18560536
- [Background] Jedrychowski W, Bendkowska I, Flak E, Penar A, Jacek R, Kaim I, Spengler JD, Camann D, Perera FP. Estimated risk for altered fetal growth resulting from exposure to fine particles during pregnancy: an epidemiologic prospective cohort study in Poland. Environ Health Perspect. 2004 Oct;112(14):1398-402. doi: 10.1289/ehp.7065. PMID 15471732
- [Background] Slama R, Thiebaugeorges O, Goua V, Aussel L, Sacco P, Bohet A, Forhan A, Ducot B, Annesi-Maesano I, Heinrich J, Magnin G, Schweitzer M, Kaminski M, Charles MA; EDEN Mother-Child Cohort Study Group. Maternal personal exposure to airborne benzene and intrauterine growth. Environ Health Perspect. 2009 Aug;117(8):1313-21. doi: 10.1289/ehp.0800465. Epub 2009 Apr 1. PMID 19672414
- [Background] Slama R, Morgenstern V, Cyrys J, Zutavern A, Herbarth O, Wichmann HE, Heinrich J; LISA Study Group. Traffic-related atmospheric pollutants levels during pregnancy and offspring's term birth weight: a study relying on a land-use regression exposure model. Environ Health Perspect. 2007 Sep;115(9):1283-92. doi: 10.1289/ehp.10047. PMID 17805417
- [Background] Lepeule J, Caini F, Bottagisi S, Galineau J, Hulin A, Marquis N, Bohet A, Siroux V, Kaminski M, Charles MA, Slama R; EDEN Mother-Child Cohort Study Group. Maternal exposure to nitrogen dioxide during pregnancy and offspring birth weight: comparison of two exposure models. Environ Health Perspect. 2010 Oct;118(10):1483-9. doi: 10.1289/ehp.0901509. Epub 2010 May 14. PMID 20472526
- [Background] Wu J, Ren C, Delfino RJ, Chung J, Wilhelm M, Ritz B. Association between local traffic-generated air pollution and preeclampsia and preterm delivery in the south coast air basin of California. Environ Health Perspect. 2009 Nov;117(11):1773-9. doi: 10.1289/ehp.0800334. Epub 2009 Jun 23. PMID 20049131
- [Background] Gulliver J, Briggs DJ. Time-space modeling of journey-time exposure to traffic-related air pollution using GIS. Environ Res. 2005 Jan;97(1):10-25. doi: 10.1016/j.envres.2004.05.002. PMID 15476729
- [Background] Cooper AR, Page AS, Wheeler BW, Hillsdon M, Griew P, Jago R. Patterns of GPS measured time outdoors after school and objective physical activity in English children: the PEACH project. Int J Behav Nutr Phys Act. 2010 Apr 22;7:31. doi: 10.1186/1479-5868-7-31. PMID 20412582
- [Background] Colquhoun DR, Goldman LR, Cole RN, Gucek M, Mansharamani M, Witter FR, Apelberg BJ, Halden RU. Global screening of human cord blood proteomes for biomarkers of toxic exposure and effect. Environ Health Perspect. 2009 May;117(5):832-8. doi: 10.1289/ehp.11816. Epub 2008 Dec 2. PMID 19478969
- [Background] Hauser R, Meeker JD, Park S, Silva MJ, Calafat AM. Temporal variability of urinary phthalate metabolite levels in men of reproductive age. Environ Health Perspect. 2004 Dec;112(17):1734-40. doi: 10.1289/ehp.7212. PMID 15579421
- [Background] de Klerk NH, English DR, Armstrong BK. A review of the effects of random measurement error on relative risk estimates in epidemiological studies. Int J Epidemiol. 1989 Sep;18(3):705-12. doi: 10.1093/ije/18.3.705. PMID 2807678
- [Background] Zanobetti A, Canner MJ, Stone PH, Schwartz J, Sher D, Eagan-Bengston E, Gates KA, Hartley LH, Suh H, Gold DR. Ambient pollution and blood pressure in cardiac rehabilitation patients. Circulation. 2004 Oct 12;110(15):2184-9. doi: 10.1161/01.CIR.0000143831.33243.D8. Epub 2004 Oct 4. PMID 15466639
- [Background] Amsallem F, Gauthier R, Ramonatxo M, Counil F, Voisin M, Denjean A, Matecki S; Groupe des EFR pediatriques, Societe Francais de Physiologie. [Respiratory function testing in infants: recommendations on normal values]. Rev Mal Respir. 2008 Apr;25(4):405-32. doi: 10.1016/s0761-8425(08)71583-3. French. PMID 18536627
- [Background] Horsley A. Lung clearance index in the assessment of airways disease. Respir Med. 2009 Jun;103(6):793-9. doi: 10.1016/j.rmed.2009.01.025. Epub 2009 Feb 25. PMID 19246184
- [Derived] Jovanovic N, Mustieles V, Althuser M, Lyon-Caen S, Alfaidy N, Thomsen C, Sakhi AK, Sabaredzovic A, Bayat S, Couturier-Tarrade A, Slama R, Philippat C. Associations between synthetic phenols, phthalates, and placental growth/function: a longitudinal cohort with exposure assessment in early pregnancy. Hum Reprod Open. 2024 Apr 1;2024(2):hoae018. doi: 10.1093/hropen/hoae018. eCollection 2024. PMID 38689737